CLINICAL TRIAL: NCT00557453
Title: The Role of Antibiotic Treatment in Patients With Acute Mild Cholecystitis - A Prospective Randomized Controlled Trial
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Dr. Haggi Mazeh, Hadassah Medical Organization
Other Study IDs: cholecystitis-HMO-CTIL
Record Dates: First submitted 2007-11-11; First posted 2007-11-14 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-04

CONDITIONS: Acute Cholecystitits

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Antibiotic treatment
  Interventions: Drug: Antibiotic treatment
- B: Non antibiotic treatment
  Interventions: Drug: No antibiotics

INTERVENTIONS:
Drug: Antibiotic treatment — Cefuroxime 750mg X3/d, Ampicillin 2G X4/d, Flagyl 500mg X3/d, Augmentin 1G X3/d, Gentamycin 240mg X1/d, Clindamycin 600mg X3/d, Ciprofloxacin 400mg X2/d All drugs will be administered IV until clinical improvement.
  Groups: A
Drug: No antibiotics — Allowed medications for both groups will include PPI / H2 blockers, home medication, SC insulin for diabetes, and SC clexane if indicated.
  Groups: B

SUMMARY:
The treatment of acute cholecystitis includes limited oral intake, antibiotics and early or delayed surgery. To date there are no randomized trials proving the benefit of antibiotic treatment.

The aim of this study is to prospectively and randomly compare between patients that are admitted for acute cholecystitis and treated with or without antibiotics.

DETAILED DESCRIPTION:
Cholelithiasis and inflammatory biliary tract disease constitute a major health problem in western countries. Acute cholecystitis is the third major cause of emergency admission to a surgical ward and its incidence increases with increasing age. Acute cholecystitis is defined as acute inflammation of the gallbladder which is commonly caused by gallstones which are impacted in the cystic duct. The treatment of acute cholecystitis varies between different medical centers around the world. In some hospitals, mainly in the US, the most common treatment is early laparoscopic cholecystectomy within 72 hours from the onset of symptoms / admission. However, in the UK and many other centers in Europe the treatment of acute cholecystitis is conservative (NPO, IV fluids and antibiotics) and laparoscopic cholecystectomy is delayed. The reasons for delayed surgery differ between institutions and include the assumption of decreased complications, surgeon and OR availability and schedule, costs, and hospital policy.

A recent metanalysis proved similar safety and efficacy of early and delayed laparoscopic cholecystectomy. The conversion rate, length of operation and complication rate (overall complication rate, intra-abdominal collection, bile leak, and CBD injury) were also comparable.

At Hadassah-Hebrew University Medical Center, Mount Scopus patients with acute cholecystitis are treated conservatively followed by delayed laparoscopic cholecystectomy. Over the years this approach proved to carry relatively low rate of complications, mainly bile duct injuries <1%, without interruption to the busy OR schedule.

Regardless to the lack of evidence based guidelines for the treatment of acute cholecystitis the traditional triad of NPO, IV fluids and antibiotics was adopted at our institution vis-à-vis the higher complication and conversion rate for early cholecystectomy. The antibiotic treatment is associated with side effects, costs and most important unavoidable development of bacterial drug resistance. However, to date there are no randomized trials proving the superiority of either one of these methods.

ELIGIBILITY:
Inclusion Criteria:

Patients with the diagnosis of mild acute cholecystitis that meet the following:

1. Sonographic (or CT) findings:

   1. cholelithiasis or sludge and
   2. wall thickening > 4 mm, and
   3. positive sonographic Murphy sign,
   4. distended gallbladder (optional)
   5. pericystic fluid (optional)
2. Additional one of the following:

   1. epigastric or RUQ pain
   2. fever > 38.0
   3. WBC > 10,000

Exclusion criteria:

1. Age - less than 18 or above 70
2. Pregnant females
3. Unconsentable patients
4. NYHA > 3
5. Use of steroids or immunosuppression
6. Onset of typical abdominal pain for over than 72 hours
7. Hemodynamic instability
8. Fever > 39 or chills
9. Palpable inflammatory RUQ mass
10. Presence of peritonitis on physical examination
11. WBC > 18,000
12. Diastase > 200 (NL 20-100)
13. Bilirubin > 85 (X5 the norm)
14. Multi organ failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted through the emergency department that are diagnosed with acute cholecystits and meet the inclusion criteria will be given the opportunity to participate in the trial. Informed consent is required. Patients may withdraw from the study at any time without giving reasons and without jeopardizing further treatment.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haggi Mazeh, M.D., Principal Investigator — Hadassah Medical Organization; Herbert R Freund, M.D., Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Yoshida M, Takada T, Kawarada Y, Tanaka A, Nimura Y, Gomi H, Hirota M, Miura F, Wada K, Mayumi T, Solomkin JS, Strasberg S, Pitt HA, Belghiti J, de Santibanes E, Fan ST, Chen MF, Belli G, Hilvano SC, Kim SW, Ker CG. Antimicrobial therapy for acute cholecystitis: Tokyo Guidelines. J Hepatobiliary Pancreat Surg. 2007;14(1):83-90. doi: 10.1007/s00534-006-1160-y. Epub 2007 Jan 30. PMID 17252301